CLINICAL TRIAL: NCT02928094
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter, Phase 3 Study to Evaluate the Safety and Efficacy of Ad5FGF-4 in Patients With Refractory Angina Due to Myocardial Ischemia
Brief Title: Ad5FGF-4 In Patients With Refractory Angina Due to Myocardial Ischemia
Acronym: AFFIRM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angionetics Inc. (Industry)
Collaborators: Huapont Life Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-3-003
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Angina, Stable
Keywords: refractory angina; myocardial ischemia; angiogenesis
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A: Ad5FGF-4 (Experimental): Ad5FGF-4, administered one time at 6x10e9 viral particles in buffer, and maximally-tolerated medical therapy for angina.
  Interventions: Biological: Ad5FGF-4
- B: Placebo (Placebo Comparator): Placebo buffer, administered one time, and maximally-tolerated medical therapy for angina.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad5FGF-4 — Ad5FGF-4 administered via intracoronary infusion using standard balloon catheter, and under conditions of transient ischemia.
  Other Names: Generx; alferminogene tadenovec
  Arms: A: Ad5FGF-4
Biological: Placebo — Placebo buffer administered via intracoronary infusion using standard balloon catheter, without transient ischemia.
  Arms: B: Placebo

SUMMARY:
The purpose of this study is to determine whether a single intracoronary infusion of an adenovirus serotype 5 virus expressing the gene for human fibroblast growth factor-4 (Ad5FGF-4) is effective in improving angina-limited exercise duration, angina functional class, frequency of angina attacks, frequency of nitroglycerin usage, and quality of life. Half of the study participants will receive Ad5FGF-4, and half will receive placebo. The primary endpoint is the change from baseline to Month 6 in Exercise Tolerance Test (ETT) duration. Long-term safety of Ad5FGF-4 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 55-75 years of age inclusive
2. Refractory angina CCS Class III or IV
3. At least 3 angina episodes per week
4. Diagnostic coronary angiogram in the past 12 months confirming the presence of coronary artery disease in patients who are not candidates for standard interventions (PCI or CABG)
5. Patients without significant and adequate reduction or relief of angina in spite of treatment with at least two functional classes of chronic anti-angina medication at the maximally tolerated dose. Functional classes of anti-angina medications include β-blockers, calcium channel blockers, nitrates, and metabolic modulators (i.e. ranolazine). Participants must have been on a stable anti-angina medication regimen for at least 4 weeks before signing the informed consent form.
6. Documented clinical evidence of inducible ischemia on stress testing within the past 6 months [e.g. nuclear perfusion imaging (stress SPECT or PET), stress ECHO, stress MRI, stress ETT (≥1 mm ST Segment depression)].
7. Maximal exercise duration of 3-8 minutes on ETT (Modified Bruce Protocol), with patient physically unable to continue due to angina or angina equivalent (e.g. exhaustion/dyspnea), or when ETT is stopped by person administering the ETT. Patient develops ≥1mm ST segment depression on each of the qualifying baseline ETT
8. Left ventricular ejection fraction (LVEF) of ≥ 30%
9. Postmenopausal female patients, women of childbearing potential and men willing to use an effective contraception method while in the study and/or who agree not to become pregnant or make their partner pregnant throughout the study and during one year after administration of the study drug
10. Female subjects of childbearing potential who have a negative urine pregnancy test and are willing to use an acceptable form of birth control during the study. For the purpose of this study, a female of childbearing potential is a female who is not postmenopausal for greater than 2 years, has not had a tubal ligation, and has not had a hysterectomy. For the purpose of this study, the following are considered acceptable methods of birth control:

    * Oral contraceptives, contraceptive patches/implants
    * Intrauterine device (IUD) together with condom or spermicide for at least three months
    * Condom and spermicide
    * Abstinence with a documented second acceptable method of birth control should the subject become sexually active
11. Willing and able to comply with all study requirements, including adherence to the assigned strategy, medical therapy, and follow-up
12. Provided written informed consent

Exclusion Criteria

1. Female patients who are pregnant, lactating (breast milk feeding), or planning a pregnancy during the course of the study and one year after administration of the study drug. Women of childbearing potential who are not using an acceptable method of birth control (i.e., IUD, oral contraceptive plus barrier contraceptive, hormone delivery system plus barrier contraceptive or condom in combination with contraceptive cream, jelly or foam). Women of childbearing potential with a positive urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) before randomization.
2. Patients with unstable angina for whom an immediate revascularization procedure (PCI or CABG) is indicated
3. Patients for whom a cardiac revascularization procedure (PCI or CABG) is planned in the next 3 months
4. Myocardial infarction within the past 3 months prior to the Screening visit
5. Congestive heart failure New York Heart Association (NYHA) Class IV
6. Myocarditis or restrictive pericarditis
7. Diagnostic coronary angiogram finding of left main coronary stenosis ≥70% (unless the patient has a patent graft or collateral vessels supplying the left coronary circulation) or proximal stenoses ≥70% in all major coronary conduit vessels (coronary arteries and bypass grafts)
8. A single patent coronary conduit (for example, totally occluded RCA and LCx with no bypass grafts. Patient will not tolerate balloon occlusion of the LAD for infusion)
9. Patients whose angiogram shows a good anatomy for angioplasty and who are candidates for that procedure. Patients without a prior angiogram or angiogram report are excluded.
10. Clinically significant aortic or mitral valvular heart disease
11. Life-threatening coronary ostial stenosis that precludes adequate catheter engagement in any target vessel, unless the vessel can be accessed via a patent bypass graft
12. Coronary artery to venous communications, which bypass the coronary capillary bed
13. Untreated life-threatening ventricular arrhythmias
14. Uncontrolled arterial hypertension with systolic blood pressure >140 mm Hg and/or diastolic pressure >100 mm Hg
15. CABG surgery within the past 6 months, unless those grafts are now occluded
16. Percutaneous coronary intervention (PCI) within the past 3 months, unless the stented/dilated vessel(s) are now occluded
17. Enhanced external counterpulsation (EECP) within 3 months prior to the start of screening evaluations
18. Prior treatment with spinal cord stimulation
19. Prior treatment with coronary sinus reducer
20. Transmyocardial or percutaneous myocardial laser revascularization within the past 12 months
21. Prior treatment with any cardiovascular gene or cell therapy within the past 12 months
22. Active SARS-CoV-2 infection (COVID-19)
23. Any major organ disease or any medical disease or condition that substantially impairs life expectancy
24. History of cancer within the past 5 years, other than basal cell carcinoma, or patients with any laboratory or physical exam or diagnostic procedure finding suggestive of current malignancy
25. Moderate to severe non-proliferative or proliferative retinopathy from any cause, clinically significant macular edema, or previous pan-retinal photocoagulation therapy
26. Heparin induced thrombocytopenia or history of idiopathic thrombocytopenic purpura or other medical condition causing thrombocytopenia
27. Serum glutamic pyruvic transaminase (SGPT) level greater than 2.0 times the upper limit of the laboratory normal range.
28. Bilirubin level ≥ 2.0 mg/dL
29. Serum creatinine ≥ 2.5 mg/dL
30. Platelet count < 100,000/μL
31. White blood cell count < 3,000/μL
32. HbA1c > 9% in patients with diabetes
33. Positive test for hepatitis B or C
34. Positive test for human immunodeficiency virus (HIV)
35. Prior anaphylaxis reaction to iodinated contrast agents
36. Patients who are known to be immunosuppressed or are receiving chronic treatment with immunosuppressive drugs
37. Received an investigational drug or biologic within 30 days of screening or are currently participating in an investigational drug, biologic or device trial
38. History of alcohol or drug abuse
39. History of non-compliance with medical therapy

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Exercise Tolerance Test (ETT) duration | Baseline and Month 6
  Modified Bruce Protocol with exercise duration limited by angina or angina equivalent

SECONDARY OUTCOMES:
Change in patient functional status (CCS class) | Baseline and Month 6
  Canadian Cardiovascular Society (CCS) angina classification
Change in weekly angina frequency | Baseline and Month 6
  Average weekly angina episodes
Change in weekly nitroglycerin usage | Baseline and Month 6
  Average weekly nitroglycerin usage
Change in quality of life | Baseline and Month 6
  Seattle Angina Questionnaire
Safety of Ad5FGF-4 | Through Month 6
  Adverse events and clinical laboratory testing
Long-term safety of Ad5FGF-4 | Through Month 60
  Occurrence of clinically significant events

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Henry TD, Grines CL, Watkins MW, Dib N, Barbeau G, Moreadith R, Andrasfay T, Engler RL. Effects of Ad5FGF-4 in patients with angina: an analysis of pooled data from the AGENT-3 and AGENT-4 trials. J Am Coll Cardiol. 2007 Sep 11;50(11):1038-46. doi: 10.1016/j.jacc.2007.06.010. Epub 2007 Aug 24. PMID 17825712
- [Background] Grines CL, Watkins MW, Mahmarian JJ, Iskandrian AE, Rade JJ, Marrott P, Pratt C, Kleiman N; Angiogene GENe Therapy (AGENT-2) Study Group. A randomized, double-blind, placebo-controlled trial of Ad5FGF-4 gene therapy and its effect on myocardial perfusion in patients with stable angina. J Am Coll Cardiol. 2003 Oct 15;42(8):1339-47. doi: 10.1016/s0735-1097(03)00988-4. PMID 14563572
- [Background] Rubanyi GM. Angiogenic gene therapy for refractory angina. Expert Opin Biol Ther. 2016;16(3):303-15. doi: 10.1517/14712598.2016.1122753. Epub 2015 Dec 14. PMID 26581236